CLINICAL TRIAL: NCT01113164
Title: Matching Genotypes and Serotonergic Medications for Alcoholism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, George Kenna, PI, Brown University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: AA016079-01A1; NCT00856128 (obsolete NCT alias)
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Alcoholism
Keywords: ondansetron; sertraline; lab studies; alcoholism; alcohol dependence
MeSH Terms: conditions — Alcoholism | interventions — Ondansetron; Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ondansetron, Placebo, Sertraline (Experimental): LL-carriers receiving ondansetron compared to either placebo or sertraline, will result in a significant reduction in alcohol consumption.
  Interventions: Drug: Ondansetron and Sertraline
- Sertraline, Placebo, Ondansetron (Experimental): SL and SS-carriers receiving sertraline compared to either placebo or ondansetron, will result in a significant reduction in alcohol consumption.
  Interventions: Drug: Ondansetron and Sertraline

INTERVENTIONS:
Drug: Ondansetron and Sertraline — capsule 0.25mg twice a day for 21 days and capsule 100mg twice a day

SUMMARY:
Sertraline, a serotonin-specific reuptake inhibitor (SSRI) that increases basal serotonin levels, was shown to reduce alcohol consumption in lower risk/severity and later onset (LOA) but not higher risk/severity earlier onset alcoholic individuals (EOA). By contrast, ondansetron, a 5-HT3 receptor reduced alcohol consumption in EOAs but not LOAs. To explain this contrast in clinical efficacy, one approach suggests that differential serotonergic response is based on a functional polymorphism of the 5-HTTLPR promoter region of the serotonin re-uptake transporter (SERT). These alleles have typically been classified as biallelic genotypes: LL, SS and SL. The LL variant is postulated to be associated with EOA and the SS/SL variants associated with LOA. To test this hypothesis the investigators therefore propose to match and mismatch serotonergic treatments to genetic polymorphic variants [in 132 non-treatment seeking alcohol dependent volunteers] in a double-blind placebo controlled 2 x 2 design human laboratory study. The investigators propose to randomize non-treatment-seeking alcohol dependent persons based on their 5'-HTTLPR variant genotype (LL or SS/SL) into one of two counterbalanced arms: participants in the first arm (LL) will first receive one drug (either 200mg/day of sertraline or ondansetron 0.5mg/day) for three weeks followed by an alcohol self-administration experiment (ASAE), [with a 1 week down-titration period if sertraline received first, during the first week of the "placebo period"] then receive placebo for two more weeks (this will be a single-blind portion to use as a comparison group and to wash out the pharmacodynamic effects of the first drug) followed by a second ASAE. Participants will then receive the second drug for three weeks followed by a third ASAE [all will receive medication for an additional 1 week period and those receiving sertraline last will be down-titrated]. Participants in the second arm (SS/SL) will receive the same medications in the same balanced design. Individuals in both arms will receive weekly medication management to enhance medication adherence. The long-term objective of this research is to prospectively examine serotonergic treatment matching for alcohol dependence based on genotyping. Of equal importance, the investigators also recognize the strong contribution of additional genetic and environmental influences on alcohol consumption.

DETAILED DESCRIPTION:
Medications and genetics have been identified as research priorities by NIAAA. The present application proposes to test two genetic-drug matching hypotheses to better understand heterogeneity among alcoholics. Previous basic science, treatment and genetic research suggests that active drinkers with the LL genetic variant of the serotonin transporter 5'-HTTLPR (a hypothesized genetic risk factor for early onset alcoholism) will respond better to ondansetron than sertraline or placebo. Conversely, active drinkers with the SS or SL genetic variant of the serotonin transporter 5'-HTTLPR (a hypothesized genetic risk factor for late onset alcoholism) will respond better to sertraline than ondansetron or placebo. The objective of this research is to match and mismatch serotonergic treatments to genetic polymorphic variants in a double-blind placebo controlled 2 x 2 design laboratory study where the 2 arms will be counterbalanced. The specific aims are to investigate: (1) whether LL-carriers receiving ondansetron results in a significant reduction in alcohol consumption during an alcohol self-administration experiment (ASAE) and during the period of treatment; (2) whether SL and SS-carriers receiving sertraline will result in a significant reduction in alcohol consumption during an ASAE and during the period of treatment; (3) examine mechanism of action for craving and subjective effects during the ASAE sessions: (4) whether there is a reduction in alcohol consumption during the ASAEs in the presence of the LG, and LA 5-HTTLPR variants and when LL participants receive ondansetron or when LL participants receive sertraline; (5) if the primary aims are moderated by the presence of the C (-1019) G polymorphism of the 5-HT1A gene promoter. We propose to randomize 132 non-treatment-seeking alcohol dependent participants based on their 5'-HTTLPR variant genotype (LL or SS/SL) into one of two counterbalanced arms: e.g. subjects in the first arm will first receive one drug (either 200mg/day of sertraline or ondansetron 0.5mg/day) for three weeks followed by an ASAE, then receive placebo for three weeks (this will be a single-blind portion to use as a comparison group and to wash out the pharmacodynamic effects of the first drug) followed by a second ASAE. Finally, participants will receive the second drug for three weeks followed by a third ASAE. Volunteers in the second arm will receive the same medications in a counter-balanced fashion. There will be a 1-week down titration after the first and third segments for all subjects. The long-term objective of this proposed research is to examine serotonergic treatment matching for alcohol dependence based on genotyping, and begin to investigate patient variation when matched prospectively with one serotonergic treatment or the other.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between 21 and 65 years old (inclusive).
2. Participants may be male or female and must be in good health as confirmed by medical history, baseline physical examination, ECG, laboratory tests, urinalysis and vital signs.
3. Female participants must be:

   Postmenopausal for at least one year, surgically sterile, or Practicing an effective method of birth control before entry and throughout the study; have a negative urine pregnancy test at baseline screening and prior to the alcohol challenge sessions.
4. Participants must understand that this is not a treatment study.
5. A diagnosis of Alcohol dependence using Module E of the structured clinical interview for the DSM-IV (SCID). Alcohol dependent as defined by an AUDIT score ≥ 12 and men must consume ≥ 35 and women ≥ 28 standardized alcoholic beverages a week.
6. Participants must be willing to take oral medication, adhere to the medication regimen and be willing to return for weekly visits and the alcohol challenge sessions.
7. Participants must be able to read and comprehend written instructions and comprehend and complete all scale and inventories required by the protocol.
8. Participants must have signed an informed consent indicating they understand the purpose of and procedures required for the study and willingness to participate.

Exclusion Criteria:

1. Pregnancy or breast feeding women.
2. Positive urine drug screen at baseline for any illegal substance other than marijuana.
3. Participants will be excluded if they have: (a) clinically significant medical abnormalities (i.e. ECG, hematological assessment, bilirubin > 150% of the upper limit of normal or ALT or AST elevations >300% the upper limit of normal, biochemistry including urinalysis, electrolytes,). (Persons with medical conditions that are adequately controlled by their primary care physician will not be excluded.)
4. Current use of psychotropic medications that cannot be discontinued
5. Medical contraindications for use of sertraline or ondansetron
6. Taking drugs that interfere with the metabolism of either drug that cannot be stopped per study physician.
7. Allergic to sertraline or ondansetron
8. Must have a breath alcohol concentration (BrAC) = 0.000 at the beginning of the alcohol challenge sessions.
9. Creatinine clearance ≤ 60 dl/min.
10. Individuals with a reasonable expectation of being institutionalized during the course of the trial or pending legal charges.
11. Participants who have significant alcohol withdrawal symptoms (clinical institute withdrawal assessment for alcohol revised (CIWA-Ar) >10.
12. lifetime depression or a history of suicide
13. history of seizures (e.g. epilepsy) or migraine headaches -

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2008-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of drinks/day consumed | 13 weeks
  To evaluate the efficacy of ondansetron for reducing drinking in participants who carry the LL variant of the serotonin transporter gene (5-HTTLPR): We hypothesize that LL-carriers receiving ondansetron compared to either placebo or sertraline, will result in a significant reduction in alcohol consumption.

SECONDARY OUTCOMES:
Number of Drinks/Day consumed. | 13 weeks
  To evaluate the efficacy of sertraline for reducing drinking in participants who carry either the SL or SS variants of the 5-HTTLPR: We hypothesize that SL and SS-carriers receiving sertraline compared to either placebo or ondansetron, will result in a significant reduction in alcohol consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

REFERENCES:
- [Background] Kenna GA, Zywiak WH, McGeary JE, Leggio L, McGeary C, Wang S, Grenga A, Swift RM. A within-group design of nontreatment seeking 5-HTTLPR genotyped alcohol-dependent subjects receiving ondansetron and sertraline. Alcohol Clin Exp Res. 2009 Feb;33(2):315-23. doi: 10.1111/j.1530-0277.2008.00835.x. Epub 2008 Nov 19. PMID 19032576
- [Derived] Kenna GA, Zywiak WH, Swift RM, McGeary JE, Clifford JS, Shoaff JR, Vuittonet C, Fricchione S, Brickley M, Beaucage K, Haass-Koffler CL, Leggio L. Ondansetron reduces naturalistic drinking in nontreatment-seeking alcohol-dependent individuals with the LL 5'-HTTLPR genotype: a laboratory study. Alcohol Clin Exp Res. 2014 Jun;38(6):1567-74. doi: 10.1111/acer.12410. Epub 2014 Apr 28. PMID 24773166